CLINICAL TRIAL: NCT02189720
Title: An Open-Label, Expanded Access Protocol for Firdapse® (Amifampridine Phosphate; 3,4-Diaminopyridine Phosphate) Treatment in Pediatric Patients With Lambert-Eaton Myasthenic Syndrome (LEMS), and in Pediatric and Adult Patients With Congenital Myasthenic Syndromes (CMSs)
Brief Title: Expanded Access Study Amifampridine Phosphate in Lambert-Eaton Myasthenic Syndrome (LEMS),Congenital Myasthenic Syndrome
Acronym: EAP-001
Status: Approved for marketing | Type: Expanded Access
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP-001
Record Dates: First submitted 2014-07-05; First posted 2014-07-15 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2024-05

CONDITIONS: Congenital Myasthenic Syndrome; Lambert-Eaton Myasthenic Syndrome; Nystagmus, Acquired
Keywords: Amifampridine Phosphate; Amifampridine; 3,4-Diaminopyridine Phosphate; 3,4-Diaminopyridine; 3,4-DAP; CMS; Congenital Myasthenic Syndrome; Neuromuscular; Expanded Access; Firdapse®; LEMS
MeSH Terms: conditions — Myasthenic Syndromes, Congenital; Lambert-Eaton Myasthenic Syndrome; Nystagmus, Pathologic | interventions — Amifampridine

INTERVENTIONS:
Drug: Amifampridine Phosphate — Dosage form: tablets containing the equivalent of 10 mg amifampridine per tablet.
  Amifampridine Phosphate given based on Investigator assessment of optimal neuromuscular benefit. In adult patients > 16 years of age, Doses ranged from 30 mg to 80 mg, divided into doses taken 3 to 4 times per day and in pediatric patients age < 16 years the maximum daily dose was 60 mg/day. No single dose to exceed 20 mg.
  Other Names: 3,4-Diaminopyridine Phosphate; 3,4 DAP; Firdapse®

SUMMARY:
Primary:

The primary objective of this study under the original protocol was to provide neuromuscular specialists and neurologists access to amifampridine phosphate therapy for their patients with LEMS, CMS or downbeat nystagmus until the product became commercially available.

Secondary:

The secondary objective of this study under the original protocol was to provide additional long-term safety data on amifampridine phosphate in patients.

Primary The primary objective of this study after its fifth amendment was to provide access to amifampridine phosphate therapy to pediatric patients with LEMS, and pediatric and adult patients with CMS until the product became commercially available for these indications or development of the product for the indication was terminated.

Secondary:

The secondary objective of this study after its fifth amendment was to assess the long-term safety of amifampridine phosphate in pediatric patients with LEMS, and pediatric and adult patients with CMS.

DETAILED DESCRIPTION:
This multicenter, expanded access study was designed to allow EAP-001 Investigators, neuromuscular specialists, and neurologists access to amifampridine phosphate therapy for their patients with LEMS, CMS, or downbeat nystagmus until such time the product became commercially available for these specific indications or development of the product for the indication was terminated. Given that these are chronic conditions, this study obtained some long-term safety data by evaluating Adverse Events, physical exams, vital signs, standard safety laboratory tests (chemistry, hematology, and urinalysis), pregnancy testing (if applicable) and abnormal ECG findings, where each of these data/measures were performed as part of a routine standard of care treatment provided by the Principal Investigator or the patient's personal physician(s) (i.e., could be performed by a different physician not involved in the treatment of neuromuscular disease).

Planned -100 sites in US and up to 200 patients. Actual- 50 sites activated and 200 patients enrolled.

Patients were seen at screening/baseline, Day 1 and at least once per year at the PIs discretion. With the COVID-19 Pandemic, telehealth visits were allowed and assessments that could be completed via remote telehealth visits were performed via phone or videoconference. Follow-up visits included Physical exams, vital signs, standard safety laboratory tests (chemistry, hematology, and urinalysis), pregnancy testing (if applicable) and ECGs.

Patients were titrated to an optimal individualized dose of amifampridine phosphate based on Principal Investigator assessment of optimal neuromuscular benefit. In patients already taking amifampridine base, amifampridine phosphate was started at an equivalent or lower dose of amifampridine phosphate, at the Principal Investigator's discretion. Therapeutic doses were to range from 10 to 80 mg, divided into doses taken two (2) to four (4) times per day, with a maximum single dose of 20 mg. For upward titration, amifampridine phosphate could be increased by 10 mg increments every four (4) to five (5) days to a maximum of 80 mg per day (ages >16 years), and to a maximum of 60 mg (ages 2 to 16 years) based on optimal neuromuscular benefit and at the discretion of the Principal Investigator. If needed, titration could occur in 5 mg/dose and per day increments. Drug was shipped to the clinic for the first dose ( Day 1) and subsequent shipments were sent to the patients home by a specialty pharmacy.

In addition to amifampridine phosphate, patients received best supportive care (BSC) treatment as determined by the Principal Investigator using concomitant medications permitted by protocol, including selected oral immunosuppressant's (i.e., prednisone or other corticosteroids, azathioprine, mycophenolate) and peripherally acting cholinesterase inhibitors (e.g., pyridostigmine). Changes to BSC could be made at the Principal Investigator's discretion, as long as prohibited concomitant medications were not used.

Firdapse® was approved for adult patients with LEMS in November 2018 and approved for pediatric patients with LEMS ages 6 years and older in September 2022. The indications for CMS and DBN were not pursued.

ELIGIBILITY:
Inclusion Criteria - Amendment 5 v6 - most recent version

* Male or female:

  * 2 years of age
* Confirmed physician diagnosis of LEMS in pediatric patients or CMS in either pediatric or adult patients.
* Completion of anti-cancer treatment at least 3 months (90 days) before treatment.
* Negative urine pregnancy test for females of childbearing potential at Screening.
* If sexually active and of childbearing potential, willing to use 2 acceptable methods of contraception from screening visit until 3 months after the last dose of investigational product. No adequate clinical data on exposed pregnancies are available for amifampridine. No nonclinical safety data are available regarding the effects of amifampridine on reproductive function. Amifampridine phosphate should not be used during pregnancy. It is unknown whether amifampridine is excreted in human breast milk. The excretion of amifampridine in milk has not been studied in animals. Amifampridine phosphate should not be used during breastfeeding.
* Any subject currently participating in study CMS 001 is immediately eligible for enrollment into study EAP-001, as long as inclusion/exclusion criteria are still met.
* Willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures.

Exclusion Criteria- Amendment 5 v6

* History of epilepsy and on medication/treatment for the same.
* CMS subtypes including slow-channel syndrome, LRP4 deficiency, plectin deficiency and acetylcholinesterase deficiency.
* Any subject with a LEMS diagnosis and ≥18 years of age.
* Known active brain metastasis. Patients with treated brain metastasis (radiotherapy and/or surgery) who have completed treatment for their brain metastasis >90 days before Screening, are neurologically stable (neurological symptoms grade <1), are on a stable dose of corticosteroids and have no evidence of new disease on magnetic resonance imaging (MRI) are eligible, provided they meet the other inclusion/exclusion criteria.
* Current use of dalfampridine (Ampyra®; 4-aminopyridine), and any form of 3,4 DAP other than the investigational product provided, such as amifampridine base and does not agree to discontinue use for the duration of the study.
* Use of guanidine hydrochloride within 7 days of starting amifampridine phosphate treatment.
* History of drug allergy to any pyridine-containing substances or any amifampridine phosphate excipients (i.e. microcrystalline cellulose, colloidal silicon dioxide or calcium stearate).
* Use of any other investigational product (other than 3,4 DAP or amifampridine phosphate) or investigational medical device within 30 days before starting treatment or requirement for any investigational agent before completion of all scheduled study assessments.
* An electrocardiogram (ECG) within 6 months before starting treatment that shows clinically significant abnormality(ies), in the opinion of the patient's personal physician for pediatric subjects <18 years of age.
* Breastfeeding or pregnant or planning to become pregnant (self or partner). Male patients with breastfeeding partners are not excluded from the study.
* Patients with end stage kidney disease on dialysis.
* Any condition that, in the view of the Principal Investigator, places the patient at risk, or patients with poor treatment compliance.

Inclusion Criteria: Protocol Amendment 1 ( first version IRB approved)

* Male or female:
* Confirmed genetic diagnosis of CMS.
* Negative urine pregnancy test for females of childbearing potential at Screening.
* If sexually active and of childbearing potential, willing to use 2 acceptable methods of contraception from screening visit until 3 months after the last dose of investigational product. No adequate clinical data on exposed pregnancies are available for amifampridine. No nonclinical safety data are available regarding the effects of amifampridine on reproductive function. Amifampridine phosphate should not be used during pregnancy. It is unknown whether amifampridine is excreted in human breast milk. The excretion of amifampridine in milk has not been studied in animals. Amifampridine phosphate should not be used during breastfeeding.
* Willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures.

Exclusion Criteria: Protocol Amendment 1 ( first version IRB approved)

* History of epilepsy and on medication/treatment for the same.
* CMS subtypes including slow-channel syndrome, LRP4 deficiency, and acetylcholinesterase deficiency.
* Current use of dalfampridine (Ampyra®; 4-aminopyridine), and any form of 3,4 DAP other than the investigational product provided, such as amifampridine base and does not agree to discontinue use for the duration of the study.
* Use of guanidine hydrochloride within 7 days of starting amifampridine phosphate treatment.
* History of drug allergy to any pyridine-containing substances or any amifampridine phosphate excipients (i.e. microcrystalline cellulose, colloidal silicon dioxide or calcium stearate).
* Use of any other investigational product (other than 3,4 DAP or amifampridine phosphate) or investigational medical device within 30 days before starting treatment or requirement for any investigational agent before completion of all scheduled study assessments.
* An electrocardiogram (ECG) within 6 months before starting treatment that shows clinically significant abnormality(ies), in the opinion of the patient's personal physician.
* Breastfeeding or pregnant or planning to become pregnant (self or partner). Male patients with breastfeeding partners are not excluded from the study.
* Any condition that, in the view of the Principal Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Perry Shieh, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States